CLINICAL TRIAL: NCT03266796
Title: Shared Decision Making in Physical Therapy: a Cross-sectional Observational Study
Status: Completed | Type: Observational
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Andrea Hausheer, cand. MScPT, BSc, Klinik Valens
Other Study IDs: Projekt ID: 2017-00848
Record Dates: First submitted 2017-08-05; First posted 2017-08-30 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Shared Decision Making

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients & Physical therapists: First consultations of peoples with musculoskeletal disorders and their physical therapists will be audiotaped. Audiotapes will be used to analyse the communication between the patients and their physicaltherapists to explore how much physical therapists involve their patients in the goal setting process, to see if there is a shared decision making existing.
  Interventions: Behavioral: goal setting process

INTERVENTIONS:
Behavioral: goal setting process — goal setting process during the first consultation

SUMMARY:
Shared decision making (SDM) is increasingly recommended in health care and reduces the unbalanced power between physical therapists and patients. There is an increased focus on communication between physical therapists and their patients during the goal setting process in current research. This study will focus on SDM in physical therapy goal setting.

The SDM Process includes a problem definition and different goal options. Good communication between physical therapists and patients during the goal setting process with an explicit agreeing on both sides regarding treatment goals and options improves patient satisfaction, treatment adherence and health outcomes.

Patients generally prefer to be actively involved in the shared decision making process. However, the preferred level of involvement of patients regarding decisions differs. Therefore, physical therapist should consider about patients' preferred level of involvement in shared decision making. Previous research observed SDM behaviours of physical therapists only in private practice settings. Research in other settings like the rehabilitation setting are recommended. It is unknown whether there are differences between settings in the SDM behaviours of physical therapists during first consultation.

DETAILED DESCRIPTION:
Background

Shared decision making (SDM) is increasingly recommended in health care and reduces the unbalanced power between physical therapists and patients. There is an increased focus on communication between physical therapists and their patients during the goal setting process in current research. This study will focus on SDM in physical therapy goal setting.

The SDM Process includes a problem definition and different goal options. Therefore, SDM may be especially important during the goal setting process in the first consultation, where a problem definition and several goal options are of interest.

An increased involvement of patients in SDM is based on clear information, empathy, two-way communication and respect for patients' beliefs and concerns. Therefore, patients are more willing to reveal information. Good communication between physical therapists and patients during the goal setting process with an explicit agreeing on both sides regarding treatment goals and options improves patient satisfaction, treatment adherence and health outcomes.

During the shared goal setting several topics should be discussed including patient's expectations and concerns, different possible goals and their pros and cons. The quality of this communication during the goal setting process can be evaluated by the OPTION Scale.

Patients generally prefer to be actively involved in the shared decision making process.

Previous research observed SDM behaviours of physical therapists, the patient's preferred level of involvement and the agreement between the patient's preferred level of involvement and the physical therapists' perception of the patient's preference during different therapy consultations in private practice settings.

Communication between physical therapists and patients may be affected by patient's self-efficacy and educational background and physical therapist's education and working experiences. These factors will therefore be evaluated in the planned study. In addition, therapists should consider patients individual preferences regarding their preferred level of involvement in the goal setting process. The control preference scale measures patients' preferred level of involvement and physical therapists' perception of this level.

It is unknown whether there are differences between settings in the SDM behaviours of physical therapists. SDM may be different in rehabilitation and private practice settings. As in private practice one physical therapist is treating the patient, there are several physical therapists treating the patient in rehabilitation setting.

ELIGIBILITY:
Inclusion Criteria:

musculoskeletal disorders First treatment German speaking

Exclusion Criteria:

n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients will be recruited. The planned sample may seem heterogenic because patients with all musculoskeletal conditions are included. However, the goal setting process is expected to be independent of diagnosis and the sample is therefore considered sufficiently homogeneous.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
OPTION scale | day 1 (e.g. "through study completion, an average of 1 year")
  The OPTION scale measures physical therapists behaviour in shared decision making. It is a measurement that evaluates the involvement of patients in shared decision making and was shown to be reliable (Elwyn et al., 2003). The OPTION scale includes items looking at communication between physical therapist and patient, especially an identified problem, patient's beliefs and concerns, different goal and treatment option and their pros and cons, patient's preferred level of involvement, possibilities for patient's to ask questions and a review of the physical therapist at the end.

SECONDARY OUTCOMES:
Control Preference Scale (CPS) | day 1 (e.g. "through study completion, an average of 1 year")
  The Control Preference Scale (CPS) measures physical therapists perception about their patient's preferences and patient's preference in SDM. The CPS is valid and reliable in healthcare decision making, easy to conduct and clinically relevant (Degner et al., 1997).

OTHER OUTCOMES:
General Self-Efficacy Scale (GSE) | day 1 (e.g. "through study completion, an average of 1 year")
  The General Self-Efficacy Scale (GSE) measures self-reported self-efficacy. The GSE is valid and Cronbach's alpha of internal reliability is between .76 and .90. Positive correlations to emotion, optimism, work satisfaction and negative correlations to depression, stress, health complaints, burnout and anxiety are examined. (Luszczynska et al., 2005) The GSE is potentially associated with SDM preference.
Characteristics of patients and physical therapists | day 1 (e.g. "through study completion, an average of 1 year")
  The following characteristics will be assessed because of their possible influence on SDM preferences.
  Patients: age, sex, previous therapy for current problem, profession Physiotherapists: age, sex, work experiences in years, education

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C. Hausheer, cand. MScPT, Principal Investigator — Klinik Valens
Locations (1):
- Kliniken Valens, Valens, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Beers E, Lee Nilsen M, Johnson JT. The Role of Patients: Shared Decision-Making. Otolaryngol Clin North Am. 2017 Aug;50(4):689-708. doi: 10.1016/j.otc.2017.03.006. Epub 2017 May 30. PMID 28571664
- [Result] Durand MA, Yen R, Barr PJ, Cochran N, Aarts J, Legare F, Reed M, James O'Malley A, Scalia P, Painchaud Guerard G, Elwyn G. Assessing medical student knowledge and attitudes about shared decision making across the curriculum: protocol for an international online survey and stakeholder analysis. BMJ Open. 2017 Jun 23;7(6):e015945. doi: 10.1136/bmjopen-2017-015945. PMID 28645974
- [Result] Dierckx K, Deveugele M, Roosen P, Devisch I. Implementation of shared decision making in physical therapy: observed level of involvement and patient preference. Phys Ther. 2013 Oct;93(10):1321-30. doi: 10.2522/ptj.20120286. Epub 2013 May 2. PMID 23641024
- [Result] Elwyn G, Edwards A, Wensing M, Hood K, Atwell C, Grol R. Shared decision making: developing the OPTION scale for measuring patient involvement. Qual Saf Health Care. 2003 Apr;12(2):93-9. doi: 10.1136/qhc.12.2.93. PMID 12679504
- [Result] Loh A, Simon D, Wills CE, Kriston L, Niebling W, Harter M. The effects of a shared decision-making intervention in primary care of depression: a cluster-randomized controlled trial. Patient Educ Couns. 2007 Aug;67(3):324-32. doi: 10.1016/j.pec.2007.03.023. Epub 2007 May 16. PMID 17509808
- [Result] Bertakis KD. The communication of information from physician to patient: a method for increasing patient retention and satisfaction. J Fam Pract. 1977 Aug;5(2):217-22. PMID 894226
- [Result] Brady TJ. The patient's role in rheumatology care. Curr Opin Rheumatol. 1998 Mar;10(2):146-51. doi: 10.1097/00002281-199803000-00011. PMID 9567211
- [Result] Roter DL, Hall JA, Merisca R, Nordstrom B, Cretin D, Svarstad B. Effectiveness of interventions to improve patient compliance: a meta-analysis. Med Care. 1998 Aug;36(8):1138-61. doi: 10.1097/00005650-199808000-00004. PMID 9708588
- [Result] Kaplan SH, Greenfield S, Ware JE Jr. Assessing the effects of physician-patient interactions on the outcomes of chronic disease. Med Care. 1989 Mar;27(3 Suppl):S110-27. doi: 10.1097/00005650-198903001-00010. PMID 2646486
- [Result] Duncan E, Best C, Hagen S. Shared decision making interventions for people with mental health conditions. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD007297. doi: 10.1002/14651858.CD007297.pub2. PMID 20091628
- [Result] Chewning B, Bylund CL, Shah B, Arora NK, Gueguen JA, Makoul G. Patient preferences for shared decisions: a systematic review. Patient Educ Couns. 2012 Jan;86(1):9-18. doi: 10.1016/j.pec.2011.02.004. Epub 2011 Apr 6. PMID 21474265
- [Result] Burton D, Blundell N, Jones M, Fraser A, Elwyn G. Shared decision-making in cardiology: do patients want it and do doctors provide it? Patient Educ Couns. 2010 Aug;80(2):173-9. doi: 10.1016/j.pec.2009.10.013. Epub 2009 Nov 30. PMID 19945818
- [Result] Weiss MC, Peters TJ. Measuring shared decision making in the consultation: a comparison of the OPTION and Informed Decision Making instruments. Patient Educ Couns. 2008 Jan;70(1):79-86. doi: 10.1016/j.pec.2007.09.001. Epub 2007 Oct 17. PMID 17942270
- [Result] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Result] Doyle C, Lennox L, Bell D. A systematic review of evidence on the links between patient experience and clinical safety and effectiveness. BMJ Open. 2013 Jan 3;3(1):e001570. doi: 10.1136/bmjopen-2012-001570. PMID 23293244
- [Result] Elwyn G, Edwards A, Mowle S, Wensing M, Wilkinson C, Kinnersley P, Grol R. Measuring the involvement of patients in shared decision-making: a systematic review of instruments. Patient Educ Couns. 2001 Apr;43(1):5-22. doi: 10.1016/s0738-3991(00)00149-x. PMID 11311834
- [Result] Luszczynska A, Scholz U, Schwarzer R. The general self-efficacy scale: multicultural validation studies. J Psychol. 2005 Sep;139(5):439-57. doi: 10.3200/JRLP.139.5.439-457. PMID 16285214